CLINICAL TRIAL: NCT06901791
Title: Assessing the Efficacy of Lactobacillus Rhamnosus LRa05 in Improving Blood Glucose and Gut Microbiota in Patients With Gestational Diabetes
Brief Title: Efficacy of Lactobacillus Rhamnosus LRa05 in Gestational Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK20250321
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: GDM
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Experimental): Participants will follow a controlled diet and exercise regimen, while also consuming the probiotic Lactobacillus rhamnosus LRa05 at a dosage of one stick per day (each stick contains 3 grams with 30 billion CFU), continuing until delivery.
  Interventions: Dietary Supplement: Conventional treatment and Probiotic
- Placebo Group (No Intervention): Participants will only receive standard treatment (diet control and exercise therapy) until delivery.

INTERVENTIONS:
Dietary Supplement: Conventional treatment and Probiotic — Participants will continuously take Lactobacillus rhamnosus LRa05 from the time of enrollment until delivery.
  Arms: Probiotic Group

SUMMARY:
This study aims to comprehensively evaluate the multifaceted impacts of Lactobacillus rhamnosus LRa05 on patients with gestational diabetes. Initially, the study will investigate the effects of LRa05 on improving patients' blood glucose levels and gut microbiota. Additionally, the study will assess the impact of this strain on patients' blood lipid levels, inflammatory markers, and body mass index (BMI). Furthermore, the study will also focus on its effects on thyroid function, vaginal microbiota, and bile acid metabolism in patients with gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Women diagnosed with gestational diabetes mellitus (GDM) at 24 weeks of gestation.

   Diagnostic criteria for GDM: Abnormal oral glucose tolerance test (OGTT) with an 82.5g glucose load during the 24th week of pregnancy (defined as meeting one or more of the following plasma glucose thresholds: fasting ≥ 5.1 mmol/L, 1-hour ≥ 10 mmol/L, or 2-hour ≥ 8.5 mmol/L).
2. Pregnant women aged 18 to 50 years.
3. Singleton pregnancy with a fetus confirmed to be structurally and chromosomally normal via ultrasound or other prenatal diagnostic methods.
4. No history of chronic diseases, including immune deficiency, hypertension, diabetes, kidney disease, or liver disease.
5. No consumption of probiotic-containing foods (e.g., yogurt, fermented foods, soybean paste) within the two weeks prior to the study.
6. Willing and able to provide written informed consent.
7. Capable of complying with the study protocol and follow-up requirements.

Exclusion Criteria:

1. Those who have taken items with similar functions to the test product in the short term, which may affect the judgment of the results.
2. Those with other endocrine diseases or currently using medications that affect blood glucose control.
3. Those with severe cardiovascular, kidney, or liver diseases.
4. Those with immunodeficiency diseases or currently using immunosuppressive agents.
5. Those with severe gastrointestinal diseases that may affect the absorption or metabolism of probiotics.
6. Those currently using other medications that may affect blood glucose control or lipid levels.
7. Those with a history of allergy to probiotics or any components of the study products.
8. Those with unhealthy lifestyle habits, such as smoking, alcohol consumption, or drug abuse.
9. Those who do not consume the test samples as required or do not follow up on time, resulting in uncertain efficacy.
10. Study participants deemed unsuitable by other researchers.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Blood glucose change | 16 weeks
  Assess and evaluate the improvement of patients' fasting blood glucose levels before the intervention begins, during the intervention, and after the intervention ends.

CONTACTS AND LOCATIONS:
Locations (1):
- Suzhou Municipal Hospital, Suzhou, Jiangsu, China